CLINICAL TRIAL: NCT07302490
Title: Comparison of the Effectiveness of Ultrasound-Guided Suprascapular Nerve Radiofrequency Ablation and Ultrasound-Guided Suprascapular Nerve Injection With Local Anesthetic and Corticosteroid in Patients With Chronic Shoulder Pain
Brief Title: Ultrasound-Guided Suprascapular Nerve RFA vs Steroid-Local Anesthetic Injection in Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nida Koçer Nazlıgül (Other)
Responsible Party: Sponsor-Investigator, Nida Koçer Nazlıgül, Physical Medicine and Rehabilitation Specialist (Sponsor-Investigator), Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSNRFA2025; 2024-KAEK-40 (Other: Ankara Etlik City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Shoulder Pain; Shoulder Impingement Syndrome; Rotator Cuff-Related Shoulder Pain; Suprascapular Nerve-Related Shoulder Pain
Keywords: Suprascapular nerve; Pulsed radiofrequency; PRF; Suprascapular nerve block; Shoulder pain; Chronic pain; Ultrasound-guided interventions; Corticosteroid injection; Local anesthetic injection; Shoulder proprioception
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Chronic Pain | interventions — Prolactin-Releasing Hormone; Anesthetics, Local; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel groups: suprascapular nerve pulsed radiofrequency (PRF) or suprascapular nerve block with local anesthetic and corticosteroid. Both interventions are administered once under ultrasound guidance. Follow-up assessments at baseline, 1 month, and 3 months will compare outcomes related to pain, functional disability, range of motion, shoulder proprioception, quality of life, and ultrasound-based measurements of supraspinatus muscle and tendon thickness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF Group (Active Comparator): Participants undergo a single-session pulsed radiofrequency (PRF) procedure applied to the suprascapular nerve under ultrasound guidance. PRF is delivered at a maximum temperature of 42°C for a total of 6 minutes. At the end of the procedure, 2 mL of 2% lidocaine is injected into the perineural area.
  Interventions: Procedure: Pulsed Radiofrequency (PRF) of the Suprascapular Nerve
- Nerve Block Group (Active Comparator): Participants receive suprascapular nerve block under ultrasound guidance consisting of 2 mL 2% lidocaine and 2 mL methylprednisolone acetate injected into the perineural area.
  Interventions: Procedure: Suprascapular Nerve Block with Local Anesthetic and Corticosteroid

INTERVENTIONS:
Procedure: Pulsed Radiofrequency (PRF) of the Suprascapular Nerve — Single-session PRF applied to the suprascapular nerve under ultrasound guidance. PRF is delivered at 42°C for 6 minutes. At the end of the procedure, 2 mL of 2% lidocaine is injected into the perineural area.
  Arms: PRF Group
Procedure: Suprascapular Nerve Block with Local Anesthetic and Corticosteroid — Injection of 2 mL 2% lidocaine and 2 mL methylprednisolone acetate into the perineural area under ultrasound guidance.
  Arms: Nerve Block Group

SUMMARY:
This study aims to compare the clinical effectiveness of two interventional treatments for chronic shoulder pain related to suprascapular nerve pathology: ultrasound-guided suprascapular nerve block and suprascapular nerve radiofrequency ablation (RFA).

A total of 104 patients with chronic shoulder pain were enrolled and assigned to one of the two treatment groups. Participants were evaluated at baseline, 1 month, and 3 months after the intervention. Outcome measures included pain intensity, functional disability, range of motion, kinesiophobia, quality of life, shoulder proprioception, and supraspinatus muscle and tendon thickness measured by ultrasound.

The primary aim of the study is to determine whether radiofrequency ablation provides more sustained pain relief and functional improvement compared with nerve block. The findings may help guide clinical decision-making in the management of chronic shoulder pain.

DETAILED DESCRIPTION:
Chronic shoulder pain is a common clinical condition that leads to functional limitation and reduced quality of life. This study aimed to compare the effectiveness of two interventional treatments in patients whose symptoms persisted despite conservative management: pulsed radiofrequency (PRF) of the suprascapular nerve under ultrasonographic guidance, and suprascapular nerve blockade with local anesthetic and corticosteroid.

Adult patients with at least 3 months of chronic shoulder pain, diagnosed with a shoulder pathology based on clinical evaluation and, when necessary, imaging, were included. Eligible participants underwent either PRF treatment or perineural injection of local anesthetic and corticosteroid. All patients were instructed in a home-based exercise program that included Codman exercises, scapular stabilization exercises, and strengthening of the internal and external rotator muscles.

All interventions were performed under real-time ultrasonographic guidance. For PRF, the suprascapular notch region was visualized, and a radiofrequency cannula was advanced toward the suprascapular nerve using an in-plane approach. Correct needle positioning was confirmed through standard sensory and motor stimulation techniques. PRF was then delivered at a maximum temperature of 42°C for a total duration of 6 minutes. At the end of the procedure, 2 mL of 2% lidocaine was administered.

In the nerve block group, a spinal needle was advanced to the perineural region using the in-plane technique. After negative aspiration, 4 mL of solution containing 2 mL of 2% lidocaine and 2 mL of methylprednisolone acetate was slowly injected, and appropriate perineural spread was confirmed sonographically.

Following each procedure, all patients were observed for at least 30 minutes and monitored for potential complications such as hematoma, infection, or neurological deficit. Mild procedural soreness was managed with ice application or simple analgesics as needed.

Participants were evaluated at baseline, at 1 month, and at 3 months post-intervention. Outcome measures included pain intensity, functional disability, range of motion, kinesiophobia, quality of life, shoulder proprioception assessed with the closed-kinematic chain angle reproduction test, and supraspinatus muscle and tendon thickness measured by ultrasonography. The primary objective was to determine whether PRF produced longer-lasting pain reduction and functional improvement compared with nerve block. Secondary objectives were to assess differences in proprioception, shoulder mobility, psychological factors related to pain, and ultrasound-based structural changes.

This study sought to comprehensively evaluate the relative effectiveness of two minimally invasive treatments for chronic shoulder pain using clinical, functional, psychological, and imaging-based outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 75 years, male or female. Presence of shoulder pain and/or mobility limitation for at least 3 months. Failure to benefit from medical treatment and exercise-based conservative therapy.

Voluntary participation and ability to provide written informed consent for enrollment in the study.

Exclusion Criteria:

Age younger than 18 years or older than 75 years. Shoulder pain caused by non-shoulder conditions such as cervical radiculopathy or myofascial pain syndrome.

Presence of severe chronic respiratory disease. History of intra-articular, peri-articular, or suprascapular nerve injection, or use of physical therapy modalities applied to the affected shoulder within the past 3 months.

Diagnosis of fibromyalgia. Presence of complex regional pain syndrome, entrapment neuropathy, or vascular disease affecting the same upper extremity.

Coagulopathy or bleeding diathesis. Presence of inflammatory or malignant disease. Severe psychiatric disorder or mental condition impairing cooperation or compliance.

Refusal to participate or inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2025-07-27 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain Intensity (VAS Score) | Baseline, 1 month and 3 months after the intervention
  Pain intensity will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 10. The primary outcome is the change in pain score from baseline to 3 months between the PRF group and the nerve block group. Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
SPADI (Shoulder Pain and Disability Index) Score | Baseline, 1 month, 3 months
  The Shoulder Pain and Disability Index (SPADI) assesses shoulder-related pain and functional limitations using a validated 13-item questionnaire. Scores range from 0 to 100, with higher scores indicating greater pain and disability. The outcome measure is the change in total SPADI score from baseline to 3 months.
SF-12 (Short Form-12 Health Survey: PCS & MCS) | Baseline, 1 month, 3 months
  The SF-12 is a validated measure of health-related quality of life that generates Physical and Mental Component Summary scores. Higher scores reflect better health status. This outcome assesses the change in SF-12 PCS and MCS scores from baseline to 3 months.
Tampa Scale for Kinesiophobia | Baseline, 1 month, 3 months
  The Tampa Scale (TSK) for Kinesiophobia evaluates fear of movement or reinjury. Scores range from 17 to 68, with higher scores indicating greater kinesiophobia. The outcome is the change in TSK score from baseline to 3 months.
Change in Shoulder Proprioception | Baseline, 1 month, 3 months
  Shoulder proprioception will be assessed using a closed-kinematic chain angle reproduction test. Participants attempt to replicate a predetermined joint angle, and the absolute error (in degrees) is recorded. The outcome measure is the change in angle reproduction error over time.
Change in Supraspinatus Muscle and Tendon Thickness | Baseline, 1 month, 3 months
  Ultrasound imaging will be used to measure supraspinatus muscle and tendon thickness. The outcome examines structural changes over time and compares differences between treatment groups.
Change in Shoulder Range of Motion | Baseline, 1 month, 3 months
  Active shoulder range of motion (flexion, abduction, internal and external rotation) will be measured using a goniometer. The outcome is the change in ROM values from baseline to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Genç, MD, Principal Investigator — Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves identifiable clinical information collected in a single-center setting, and current institutional and national data protection regulations do not allow the external distribution of patient-level datasets. Only aggregated results will be available upon reasonable request.